CLINICAL TRIAL: NCT01946373
Title: A Phase I Study to Evaluate Safety, Feasibility and Immunologic Response of Adoptive T Cell Transfer With or Without Dendritic Cell Vaccination in Patients With Metastatic Melanoma
Brief Title: T Cell Transfer With or Without Dendritic Cell Vaccination in Patients With Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Maria Wolodarski, Dr, Karolinska University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAT-02; 2012-000450-63 (EudraCT Number)
Record Dates: First submitted 2013-09-12; First posted 2013-09-19 (Estimated); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Melanoma
Keywords: Melanoma; Dendritic cell vaccination; Lymphodepletion; Adoptive cell transfer; T cells; Tumor infiltrating lymphocytes; Fludarabine; IL-2; Interleukin-2; Cyclophosphamide; Phase I study; Monocytes; Autologous; NY-ESO-1
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy + T cells + IL-2 (Experimental): Cyclophosphamide 60 mg/kg/d by vein (IV) daily for 2 days followed by fludarabine 25 mg/m^2 IV daily for 5 days before T cell infusion. The day after chemotherapy up to 5 x 10^10 T cells IV infusion. Interleukin-2 90 minutes after T cell infusion at a dose of 100,000 IU/kg as IV bolus over 15 minute period every 8-hours for up to 14 doses.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: T cells; Biological: Interleukin-2
- Chemotherapy + T cells + IL-2 + DCV (Experimental): Cyclophosphamide 60 mg/kg/d by vein (IV) daily for 2 days followed by fludarabine 25 mg/m^2 IV daily for 5 days before T cell infusion. The day after chemotherapy up to 5 x 10^10 T cells IV infusion. Interleukin-2 90 minutes after T cell infusion at a dose of 100,000 IU/kg as IV bolus over 15 minute period every 8-hours for up to 14 doses. After completion of the IL-2 treatment 3-5 doses of weekly intradermal vaccinations with up to 1.5 x 10^7 Dendritic cells pulsed with autologous tumor lysate and NY-ESO-1 peptide.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: T cells; Biological: Interleukin-2; Biological: Dendritic cell vaccine

INTERVENTIONS:
Drug: Cyclophosphamide
  Other Names: Sendoxan; Cytoxan; Neosar
Drug: Fludarabine
  Other Names: Fludarabine phosphate; Fludara
Biological: T cells
Biological: Interleukin-2
  Other Names: IL-2; Proleukin
Biological: Dendritic cell vaccine
  Arms: Chemotherapy + T cells + IL-2 + DCV

SUMMARY:
The purpose of this study is to learn if dendritic cell vaccine will increase the effect of tumor infiltrating lymphocytes given with chemotherapy and interleukin-2 in patients with melanoma.

DETAILED DESCRIPTION:
The MAT02 clinical trial is a phase 1 clinical trial with the objective to assess the safety, feasibility and immunological efficacy of the combined application of two immunological treatment modalities in patients with metastatic melanoma:

1. Cohort A: After a non-myeloablative conditioning regimen, 5 patients will receive one bulk infusion of T cells. T cells will be expanded ex vivo from autologous tumor infiltrating lymphocytes (TIL). In vivo persistence of the infused cells will be supported by administration of IL-2, a T cell survival factor.
2. Cohort B: This adoptive cell transfer (ACT) step will in additional 10 patients be followed by a vaccination with autologous, in vitro-generated, dendritic cells (DC), loaded with autologous tumor lysate and a synthetically produced peptide derived from the tumor associated antigen NY-ESO 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable (direct on body surface or by x-ray and/or CT) malignant melanoma (including uveal melanoma), that is advanced, inoperable stage III (advanced regional lymph node metastases, or more than 5 in-transit metastases, N2) or stage IV (distant metastasis, M1) according to the AJCC classification and confirmed by histology/cytology and appropriate radiological investigations.
* Patients with a palpable resectable lesion located in the skin or in a lymph node or a lesion accessible by (core) biopsy.
* Disease should be in progression and the patient should have exhausted other approved therapeutic options, if not the physician considers that an earlier study entry benefits the patient.
* Ambulatory performance status (ECOG 0, 1, 2).
* Age 18-74 and life expectancy greater than 3 months.

Exclusion Criteria:

* Any of the above criteria are not met.
* Significant history or current evidence of cardiovascular disease (e.g. uncontrolled congestive heart failure or hypertension, unstable coronary artery disease or serious arrhythmias) or major respiratory diseases. In questionable cases, a stress test should be performed.
* Recipients of a major organ allograft. Autoimmune diseases such as, but not limited to, inflammatory bowel disease or multiple sclerosis. Vitiligo is not an exclusion criterion. Other serious chronic diseases.
* Other serious illnesses, e.g. active infections requiring antibiotics, bleeding disorders.
* Has had prior systemic cancer therapy within the past four weeks at the time of the start of the lymphodepletion regimen.
* Patients diagnosed with prior malignancies (except adequately treated basal cell carcinomas of the skin or in situ carcinomas of the skin or in situ carcinomas of the cervix, surgically cured) within the past 5 years.
* Patients with second advanced malignancies concurrently.
* Active CNS metastases. (Note: Patients with brain metastases that have been completely resected at least one month prior to registration or have undergone gamma knife treatment with no evidence of recurrence on CT and who are neurologically stable, are not excluded).
* Organic brain syndrome or significant psychiatric disorder which would preclude participation in the full protocol and follow-up.
* Immunodeficiency, previous splenectomy or radiation therapy of the spleen.
* Screening laboratory values:

  a) Inadequate hematologic function defined by: i) White blood count (WBC) <3.0 x 109/l ii) Platelet count <100x109/l iii) Hemoglobin level <100 g/l b) Inadequate hepatic function as defined by either: i) Total bilirubin level >1.5 times the upper limit of normal (ULN) ii) Aspartate amino transferase (AST) or alanine amino transferase (ALT) >3 times the ULN (if related to liver metastases >5 times the ULN) c) Inadequate renal function defined as serum creatinine >1.5 times the ULN
* Infectious diseases that can be transmitted via contact with blood, such as HIV, Hepatitis B and C.
* Women who are pregnant or nursing will be excluded because of the potentially dangerous effects of the preparative chemotherapy on the fetus.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety of the T cell therapy, with and without dendritic cell vaccine, as evaluated according to the NCI CTCAE scale version 4.0 | 30 days

SECONDARY OUTCOMES:
Time to disease progression assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maria Wolodarski, MD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden